CLINICAL TRIAL: NCT02920632
Title: COGTIPS (COGnitive Training In Parkinson Study): The Effect of Online Cognitive Training on Cognition and Brain Networks in Parkinson's Disease
Brief Title: Cognitive Training in Parkinson Study
Acronym: cogtips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dutch Parkinson Patient Association (Other)
Responsible Party: Principal Investigator, Chris Vriend, PhD, Principle Investigator, Postdoctoral Researcher, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWO/16-10
Record Dates: First submitted 2016-08-30; First posted 2016-09-30 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; Impaired Cognition; Alteration in Cognition
Keywords: Parkinson; Cognitive training; Cognitive rehabilitation; Brain networks
MeSH Terms: conditions — Parkinson Disease; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online cognitive training 1 (Experimental): Eight-week, three times a week during 45 minutes cognitive training
  Interventions: Behavioral: Online cognitive training 1
- Online cognitive training 2 (Active Comparator): Eight-week, three times a week during 45 minutes cognitive activities
  Interventions: Behavioral: Online cognitive training 2
- Healthy control subjects (No Intervention): Reference group to compare cognitive training effects to

INTERVENTIONS:
Behavioral: Online cognitive training 1 — Eight-week online cognitive training program, three times a week for 45 minutes. The training contains several games that are designed to train cognitive functions.
  Arms: Online cognitive training 1
Behavioral: Online cognitive training 2 — Eight-week online active comparator program, three times a week for 45 minutes. The training contains several games.
  Arms: Online cognitive training 2

SUMMARY:
This study evaluates the efficacy of an eight-week online cognitive training program on objective and subjective cognitive functions in Parkinson's disease. Moreover, we intend to map the effect on brain network function, and if cognitive training can prevent the development of PD-MCI/PD-D after one- and two-year follow-up. In this study, two training groups will be compared (N: 70 vs 70). In a part of the participants MRI will be assessed (N: 40 vs. 40). We expect cognitive training to improve cognitive functions, and to improve the efficiency of brain network function. Moreover, we expect that cognitive training can decrease the risk of PD-MCI/PD-D at one- and two-year follow-up.

DETAILED DESCRIPTION:
BACKGROUND In Parkinson's disease (PD), cognitive dysfunction is frequently reported - approximately 50% of PD patients experience cognitive impairment (Litvan et al., 2011). Of these impairments, executive dysfunction is most frequently reported early in the disease trajectory (Bosboom, Stoffers, & Wolters, 2004; Muslimovic, Post, Speelman, & Schmand, 2005), while impairments in other cognitive domains (i.e. attention, episodic memory, visuospatial functions) are also highly prevalent (Bosboom et al., 2004). The majority of PD patients ultimately develops PD dementia (PD-D; Aarsland, Andersen, Larsen, Lolk, & Kragh-Sorensen, 2003; Hely, Reid, Adena, Halliday, & Morris, 2008). Moreover, about 10% of the PD patients develops PD-D every year (Aarsland & Kurz, 2010). Cognitive dysfunctions in PD have a significant negative influence on the quality of life (Klepac, Trkulja, Relja, & Babic, 2008), while treatment of these dysfunctions is in its infancy.

Cognitive training may provide a new intervention for reducing cognitive complaints and delaying the onset of mild cognitive impairment (MCI) or PD-D. This intervention has been widely studied in other diseases (Cicerone et al., 2011; Olazaran et al., 2010). Moreover, studies have provided evidence not only for behavioral influences, but also for brain connectivity and activity effects of cognitive training (Chapman et al., 2015; Castellanos et al., 2010; Subramaniam et al., 2012; Subramaniam et al., 2014; Belleville et al., 2011; Rosen, Sugiura, Kramer, Whitfield-Gabrieli, & Gabrieli, 2011). This suggests a restorative effect of cognitive training on disrupted brain networks.

In PD, cognitive dysfunction - mainly executive dysfunction - is associated with disruption of the cortico-striato-thalamo-corticale circuits by depletion of dopamine. Dysfunction of these circuits seems to disrupt several cognitive networks, which leads to cognitive dysfunction (Baggio et al., 2014). Cognitive training could counteract these disruptions by normalising activity and connectivity, and ultimately lead to a reduction of impairment. Since earlier studies in different patient populations have shown that cognitive training has lasting effects (Petrelli et al., 2015), normalising disruptions underlying cognitive impairment could prevent cognitive deterioration and therefore prevent or delay the development of PD-D.

Few studies in PD have focused on cognitive training and its neural correlates. A meta-analysis by Leung et al. (2015) showed positive effects of cognitive training on mainly 'frontal' cognitive functions (i.e. working memory, executive functions, processing speed). In addition, earlier research has described a neuroprotective effect of cognitive training on the development of MCI in PD (odds ratio: 3; Petrelli et al., 2015). Until now, however, studies have been relatively small and mainly without a controlled design - consequently, there is a need for large randomized controlled studies (Hindle, Petrelli, Clare, & Kalbe, 2013; Leung et al., 2015). Moreover, neural effects of cognitive training are largely unknown in PD. Furthermore, it is important to study the improvement of patients on daily functioning after cognitive training, rather than solely focusing on cognitive tasks and neural measures. Finally, cognitive training has been performed mainly in hospital settings, while PD patients have mobility problems - a training method suitable to perform from home is therefore needed for this population.

OBJECTIVES The study objective is primarily to measure the effect of an online cognitive training in patients with mild cognitive complaints in PD. An online training, specifically altered for PD patients (BrainGymmer) will be compared with an active comparator. In both conditions, participants will train eight weeks, three times a week during 45 minutes.

Primary objective:

- To measure the effect of an online cognitive training (as compared to the active comparator), eight weeks, three times a week, on executive functions in patients with mild cognitive complaints in PD.

Secondary objectives:

* To measure the effect of online cognitive training on daily functioning.
* To measure the endurance of the training effect after six months, one and two years.
* To assess the reduced risk of MCI and PD-D development by cognitive training.
* To assess the effect of cognitive training on brain network efficiency and connectivity.
* To assess the effect of cognitive training on brain network topology and connectivity, and cognition, relative to those of matched healthy control participants.
* To assess the difference in brain network topology and connectivity, and cognition, between Parkinson's disease patients with or without cognitive impairment and healthy control participants.

ELIGIBILITY:
--- Parkinson's disease patients ---

Inclusion Criteria:

* Subjective cognitive complaints, measured by the Parkinson's Disease Cognitive Functional Rating Scale score > 3 (PD-CFRS). A score above 3 indicates significant cognitive complaints, that are milder than complaints associated with Parkinson's disease dementia. This questionnaire is filled in by the patient.
* Participants' Hoehn & Yahr stage is lower than 4. Patients are stable on dopaminergic medication at least a month before starting the intervention. During the intervention, patient and neurologist will be asked to keep the dopaminergic medication dosage as stable as possible.
* Participants have access to a computer or tablet, with access to the Internet. If the participant uses a computer, he or she is capable of using a keyboard and computer mouse.
* Participants are willing to sign informed consent.

Exclusion Criteria:

General criteria:

* Indications for a dementia syndrome, measured by the Self-administered Gerocognitive Examination score < 14 or the Montreal Cognitive Assessment score < 22.
* Current drug- or alcohol abuse, measured by a score > 1 on the four CAGE AID-questions (according to the Trimbos guidelines).
* The inability to undergo extensive neuropsychological assessment, or eight weeks of intervention.
* Moderate to severe depressive symptoms, as defined by the Beck Depression Inventory score > 18.
* An impulse control disorder, including internet addiction, screened by the impulse control disorder criteria interview.
* Psychotic symptoms, screened by the Questionnaire for Psychotic Experiences. Benign hallucinations with insight are not contraindicated.
* Traumatic brain injury, only in case of a contusio cerebri with 1) loss of consciousness for > 15 minutes and 2) posttraumatic amnesia > 1 hour.
* A space occupying lesion defined by a radiologist, or significant vascular abnormalities (Fazekas > 1).

For participation in MRI research:

* Severe claustrophobia
* Metal in the body (for example, deep brain stimulator or pacemaker)
* Pregnancy
* Problems with or shortness of breath during 60 minutes of lying still.

  * Healthy control subjects ---

Inclusion criteria:

- Participants are willing to sign informed consent.

Exclusion criteria:

* Indications for a neurological disease, such as Parkinson's disease, Alzheimer's disease, mild cognitive impairment, multiple sclerosis or Huntington's disease;
* Indications for a dementia syndrome, measured by the Montreal Cognitive Assessment score < 22.
* Indications for a current stroke or CVA, or in the past.
* Indications for the presence of a psychotic or depressive disorder, measured with a positive screening on the SAPS-PD (benign hallucinations with insight are not contraindicated) and a BDI > 18 respectively.
* Current drug- or alcohol abuse, measured by a score > 1 on the four CAGE AID-questions (according to the Trimbos guidelines).
* The inability to undergo extensive neuropsychological assessment, or eight weeks of intervention.
* Traumatic brain injury, only in case of a contusio cerebri with 1) loss of conciousness for > 15 minutes and 2) posttraumatic amnesia > 1 hour.
* A space occupying lesion defined by a radiologist, or significant vascular abnormalities (Fazekas > 1).
* Contra-indications for participation in MRI scanning (see above)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Vriend, PhD., Principal Investigator — Amsterdam UMC, location VUmc; Odile A Van den Heuvel, MD PhD., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litvan I, Aarsland D, Adler CH, Goldman JG, Kulisevsky J, Mollenhauer B, Rodriguez-Oroz MC, Troster AI, Weintraub D. MDS Task Force on mild cognitive impairment in Parkinson's disease: critical review of PD-MCI. Mov Disord. 2011 Aug 15;26(10):1814-24. doi: 10.1002/mds.23823. Epub 2011 Jun 9. PMID 21661055
- [Background] Bosboom JL, Stoffers D, Wolters ECh. Cognitive dysfunction and dementia in Parkinson's disease. J Neural Transm (Vienna). 2004 Oct;111(10-11):1303-15. doi: 10.1007/s00702-004-0168-1. Epub 2004 Jun 30. PMID 15480840
- [Background] Muslimovic D, Post B, Speelman JD, Schmand B. Cognitive profile of patients with newly diagnosed Parkinson disease. Neurology. 2005 Oct 25;65(8):1239-45. doi: 10.1212/01.wnl.0000180516.69442.95. PMID 16247051
- [Background] Aarsland D, Andersen K, Larsen JP, Lolk A, Kragh-Sorensen P. Prevalence and characteristics of dementia in Parkinson disease: an 8-year prospective study. Arch Neurol. 2003 Mar;60(3):387-92. doi: 10.1001/archneur.60.3.387. PMID 12633150
- [Background] Hely MA, Reid WG, Adena MA, Halliday GM, Morris JG. The Sydney multicenter study of Parkinson's disease: the inevitability of dementia at 20 years. Mov Disord. 2008 Apr 30;23(6):837-44. doi: 10.1002/mds.21956. PMID 18307261
- [Background] Aarsland D, Kurz MW. The epidemiology of dementia associated with Parkinson disease. J Neurol Sci. 2010 Feb 15;289(1-2):18-22. doi: 10.1016/j.jns.2009.08.034. Epub 2009 Sep 4. PMID 19733364
- [Background] Klepac N, Trkulja V, Relja M, Babic T. Is quality of life in non-demented Parkinson's disease patients related to cognitive performance? A clinic-based cross-sectional study. Eur J Neurol. 2008 Feb;15(2):128-33. doi: 10.1111/j.1468-1331.2007.02011.x. PMID 18217883
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Olazaran J, Reisberg B, Clare L, Cruz I, Pena-Casanova J, Del Ser T, Woods B, Beck C, Auer S, Lai C, Spector A, Fazio S, Bond J, Kivipelto M, Brodaty H, Rojo JM, Collins H, Teri L, Mittelman M, Orrell M, Feldman HH, Muniz R. Nonpharmacological therapies in Alzheimer's disease: a systematic review of efficacy. Dement Geriatr Cogn Disord. 2010;30(2):161-78. doi: 10.1159/000316119. Epub 2010 Sep 10. PMID 20838046
- [Background] Chapman SB, Aslan S, Spence JS, Hart JJ Jr, Bartz EK, Didehbani N, Keebler MW, Gardner CM, Strain JF, DeFina LF, Lu H. Neural mechanisms of brain plasticity with complex cognitive training in healthy seniors. Cereb Cortex. 2015 Feb;25(2):396-405. doi: 10.1093/cercor/bht234. Epub 2013 Aug 28. PMID 23985135
- [Background] Castellanos NP, Paul N, Ordonez VE, Demuynck O, Bajo R, Campo P, Bilbao A, Ortiz T, del-Pozo F, Maestu F. Reorganization of functional connectivity as a correlate of cognitive recovery in acquired brain injury. Brain. 2010 Aug;133(Pt 8):2365-81. doi: 10.1093/brain/awq174. PMID 20826433
- [Background] Subramaniam K, Luks TL, Fisher M, Simpson GV, Nagarajan S, Vinogradov S. Computerized cognitive training restores neural activity within the reality monitoring network in schizophrenia. Neuron. 2012 Feb 23;73(4):842-53. doi: 10.1016/j.neuron.2011.12.024. PMID 22365555
- [Background] Subramaniam K, Luks TL, Garrett C, Chung C, Fisher M, Nagarajan S, Vinogradov S. Intensive cognitive training in schizophrenia enhances working memory and associated prefrontal cortical efficiency in a manner that drives long-term functional gains. Neuroimage. 2014 Oct 1;99:281-92. doi: 10.1016/j.neuroimage.2014.05.057. Epub 2014 May 24. PMID 24867353
- [Background] Belleville S, Clement F, Mellah S, Gilbert B, Fontaine F, Gauthier S. Training-related brain plasticity in subjects at risk of developing Alzheimer's disease. Brain. 2011 Jun;134(Pt 6):1623-34. doi: 10.1093/brain/awr037. Epub 2011 Mar 22. PMID 21427462
- [Background] Rosen AC, Sugiura L, Kramer JH, Whitfield-Gabrieli S, Gabrieli JD. Cognitive training changes hippocampal function in mild cognitive impairment: a pilot study. J Alzheimers Dis. 2011;26 Suppl 3(Suppl 3):349-57. doi: 10.3233/JAD-2011-0009. PMID 21971474
- [Background] Baggio HC, Sala-Llonch R, Segura B, Marti MJ, Valldeoriola F, Compta Y, Tolosa E, Junque C. Functional brain networks and cognitive deficits in Parkinson's disease. Hum Brain Mapp. 2014 Sep;35(9):4620-34. doi: 10.1002/hbm.22499. Epub 2014 Mar 17. PMID 24639411
- [Background] Petrelli A, Kaesberg S, Barbe MT, Timmermann L, Rosen JB, Fink GR, Kessler J, Kalbe E. Cognitive training in Parkinson's disease reduces cognitive decline in the long term. Eur J Neurol. 2015 Apr;22(4):640-7. doi: 10.1111/ene.12621. Epub 2014 Dec 22. PMID 25534579
- [Background] Leung IH, Walton CC, Hallock H, Lewis SJ, Valenzuela M, Lampit A. Cognitive training in Parkinson disease: A systematic review and meta-analysis. Neurology. 2015 Nov 24;85(21):1843-51. doi: 10.1212/WNL.0000000000002145. Epub 2015 Oct 30. PMID 26519540
- [Background] Hindle JV, Petrelli A, Clare L, Kalbe E. Nonpharmacological enhancement of cognitive function in Parkinson's disease: a systematic review. Mov Disord. 2013 Jul;28(8):1034-49. doi: 10.1002/mds.25377. Epub 2013 Feb 20. PMID 23426759
- [Derived] van Balkom TD, Berendse HW, van der Werf YD, Twisk JWR, Zijlstra I, Hagen RH, Berk T, Vriend C, van den Heuvel OA. COGTIPS: a double-blind randomized active controlled trial protocol to study the effect of home-based, online cognitive training on cognition and brain networks in Parkinson's disease. BMC Neurol. 2019 Jul 31;19(1):179. doi: 10.1186/s12883-019-1403-6. PMID 31366395
- See also: COGTIPS methodology article — https://doi.org/10.1186/s12883-019-1403-6
- See also: COGTIPS primary endpoint preprint/publication — https://doi.org/10.1101/2021.03.04.21252499
- See also: COGTIPS DWI results article — https://doi.org/10.1007/s13311-021-01103-9

RESULTS

PARTICIPANT FLOW:
Groups:
- Online Cognitive Training 1 (N=68): Eight-week, three times a week during 45 minutes cognitive training
  Online cognitive training 1: Eight-week online cognitive training program, three times a week for 45 minutes. The training contains several games that are designed to train cognitive functions.
- Online Cognitive Training 2 (N=68): Eight-week, three times a week during 45 minutes cognitive activities
  Online cognitive training 2: Eight-week online active comparator program, three times a week for 45 minutes. The training contains several games.
- Healthy Control Subjects (N=31): Reference group to compare cognitive training effects to
Period: Overall Study
Arm/Group | Online Cognitive Training 1 (N=68) | Online Cognitive Training 2 (N=68) | Healthy Control Subjects (N=31)
Started | 68 | 68 | 31
T1 (After Training) | 67 | 66 | 0 (not applicable: only baseline assessment visit in healthy control group)
T2 (6-mnth FU) | 64 | 62 | 0 (not applicable: only baseline assessment visit in healthy control group)
T3 (1-y FU) | 56 | 53 | 0 (not applicable: only baseline assessment visit in healthy control group)
Completed | 52 | 51 | 29
Not Completed | 16 | 17 | 2

BASELINE CHARACTERISTICS:
Population: Two healthy control subjects started participation but withdrew during MRI scanning due to in-scanner panic attacks.
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Cognitive Training 1 (N=68) | Online Cognitive Training 2 (N=68) | Healthy Control Subjects (N=31) | Total
Number analyzed (Participants) | 68 | 68 | 29 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.1) | 62.9 (7.0) | 62.3 (9.8) | 62.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 21 | 12 | 66
  Male | 35 | 47 | 17 | 99
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Unified PD Rating Scale-III - motor score (UPDRS-III) [Mean (Standard Deviation); unit: units on the motor score scale] — UPDRS-III motor score measures severity of PD motor symptoms on a continuous scale (range 0-108, higher is considered worse) Population: UPDRS-III not taken in healthy controls (disease-specific measure)
  units on the motor score scale
    number analyzed (Participants) | 68 | 68 | 0 | 136
    (all) | 20.2 (8.3) | 21.0 (9.5) |  | 20.6 (8.9)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on the MoCA scale] — MoCA measures global cognitive function on a continuous scale (range 0-30, higher is considered better)
  units on the MoCA scale | 26.3 (2.0) | 25.9 (2.3) | 28.2 (1.5) | 26.5 (2.2)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on the BDI scale] — BDI measures severity of depressive symptoms on a continuous scale (range 0-63, higher is considered worse)
  units on the BDI scale | 8.2 (4.0) | 7.9 (4.1) | 4.3 (4.2) | 7.3 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy on the Tower of London Task
Description: Change in executive function after eight weeks of cognitive training as measured by percentage correct on the Tower of London task. Accuracy is measured in percentage correct (%, range 0-100, higher is considered better).
Time Frame: Baseline (T0, "Pre-intervention") to eight weeks (T1, "Post-intervention")
Population: Number analyzed lower due to difficulty understanding the task, or no follow-up assessment in PD group and difficulty understanding the task (n=1) in healthy control group. Healthy control subjects did not undergo an intervention and T1 measurement and scores at T1 are therefore not supplied for this subgroup.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2 | Healthy Control Subjects
Number analyzed (Participants) | 62 | 64 | 28
percentage of correct responses
  Baseline - T0 | 81.2 (9.1) | 82.3 (7.9) | 88.1 (5.8)
  eight weeks - T1: number analyzed (Participants) | 62 | 64 | 0
  eight weeks - T1 | 84.0 (10.4) | 84.9 (8.2) |

2. Secondary Outcome: Total Score on Parkinson's Disease Cognitive Functional Rating Scale
Description: Score on subjective cognitive complaints after eight weeks of cognitive training, measured with the Parkinson's disease Cognitive Functional Rating Scale (PD-CFRS), with score range [0-24], where higher scores indicate more severe subjective cognitive complaints.
Time Frame: Baseline (T0, "Pre-intervention") to eight weeks (T1, "Post-intervention")
Population: Questionnaire not taken in healthy control group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2
Number analyzed (Participants) | 68 | 68
score on a scale
  Baseline - T0 | 8.0 (4.0) | 9.7 (4.7)
  Eight week - T1 | 6.9 (4.3) | 8.0 (5.1)

3. Secondary Outcome: Total Score on Cognitive Failures Questionnaire
Description: Score on subjective cognitive complaints after eight weeks of cognitive training (T0 to T1), measured by the Cognitive failures questionnaire (CFQ), a questionnaire with range [0-100] where a higher score indicates more severe subjective cognitive complaints.
Time Frame: Baseline (T0, "Pre-intervention") to eight weeks (T1, "Post-intervention")
Population: One participant in Online cognitive training 1 did not fill out the questionnaires.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2
Number analyzed (Participants) | 67 | 68
scores on a scale
  Baseline - T0 | 38.2 (10.6) | 38.5 (11.5)
  Eight week - T1 | 36.9 (10.5) | 38.0 (12.7)

4. Secondary Outcome: Reaction Time on the Tower of London Task
Description: Change on Executive function from T0 to T1, measured with the average reaction time on the Tower of London task over all trials. Reaction time is measured in seconds, where higher reaction time is considered worse.
Time Frame: Baseline (T0, "Pre-intervention") to eight weeks (T1, "Post-intervention")
Population: Number analyzed lower due to difficulty understanding the task (n=7), or no follow-up assessment (n=3) in PD group and difficulty understanding the task (n=1) in healthy control group. Healthy control subjects did not undergo an intervention and T1 measurement and scores at post-intervention are therefore not supplied.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2 | Healthy Control Subjects
Number analyzed (Participants) | 62 | 64 | 28
seconds
  Baseline - T0 | 12.4 (3.2) | 12.7 (2.7) | 11.2 (2.2)
  Eight weeks - T1: number analyzed (Participants) | 62 | 64 | 0
  Eight weeks - T1 | 11.4 (2.9) | 12.1 (2.9) |

5. Secondary Outcome: Performance on the Controlled Oral Word Association Test
Description: Executive functions CHANGE after eight weeks of cognitive training (T0 to T1), measured with the Controlled Oral Word Association Test (Letter fluency). Minimum score: 0, there is no maximum score. A higher score indicates better performance.
Time Frame: Baseline (T0, "Pre-intervention") to eight weeks (T1, "Post-intervention")
Population: Three participants dropped out of the study and did not perform the T1 measurement and were subsequently removed from analyses. Healthy control subjects did not perform the second assessment.
Measure: Mean (Standard Deviation); unit: total number of words produced
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2 | Healthy Control Subjects
Number analyzed (Participants) | 67 | 66 | 29
total number of words produced
  Baseline (T0) | 38.0 (10.6) | 38.8 (11.9) | 43.7 (9.7)
  Eight weeks (T1): number analyzed (Participants) | 67 | 66 | 0
  Eight weeks (T1) | 42.5 (12.7) | 42.6 (12.5) |

6. Secondary Outcome: Performance on Tower of London Accuracy at Six-months Follow-up
Description: Persistence of cognitive training effect on executive functions measured with the accuracy on the Tower of London task six-month after completion of the intervention. Accuracy is measured with mean percentage correct over 100 trials, where a higher percentage correct reflects better cognitive function.
Time Frame: Six months after training completion (T2)
Population: Healthy control subjects did not undergo follow-up assessment. Number of participants analyzed lower than total population due to drop-out at T2 (n=8) and difficulty understanding the task at one of the time-points (n=11)
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Online Cognitive Training 1 (N=68) | Online Cognitive Training 2 (N=68)
Number analyzed (Participants) | 57 | 60
percentage of correct responses | 84.3 (10.4) | 84.5 (9.1)

7. Secondary Outcome: Performance on Tower of London Accuracy at One-year Follow-up
Description: Persistence of cognitive training effect on executive functions measured with the accuracy on the Tower of London task one year after completion of the intervention. Accuracy is measured with mean percentage correct over 100 trials, where a higher percentage correct reflects better cognitive function.
Time Frame: One year after completion of intervention (T3, "Follow-up 2")
Population: Healthy control subjects did not undergo follow-up assessments. Number of participants analyzed differs from total sample due to drop-out (n=12), missed assessment (n=15) and difficulty understanding the task (n=2).
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2
Number analyzed (Participants) | 55 | 52
percentage of correct responses | 83.3 (14.0) | 84.7 (10.5)

8. Secondary Outcome: Performance on Tower of London Accuracy at Two-year Follow-up
Description: Persistence of cognitive training effect on executive functions measured with the accuracy on the Tower of London task two year after completion of the intervention. Accuracy is measured with mean percentage correct over 100 trials, where a higher percentage correct reflects better cognitive function.
Time Frame: Two years after completion of the intervention (T4)
Population: Healthy control subjects did not undergo follow-up assessemnts. Number of participants analyzed differs from total sample due to drop-out (n=12), missed assessment (n=21) and difficulty understanding the task.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Online Cognitive Training 1 (N=68) | Online Cognitive Training 2 (N=68)
Number analyzed (Participants) | 50 | 49
percentage of correct responses | 82.7 (11.7) | 82.1 (10.6)

9. Secondary Outcome: Conversion to Mild Cognitive Impairment or Dementia at One-year Follow-up
Description: Incidence of conversion of cognitive status at one-year follow-up with respect to the cognitive status at baseline (T0). Cognitive status is defined as cognitively normal (NC), mild cognitive impairment (MCI, according to cognitive aspects of level II MDS criteria), or dementia (according to cognitive aspects of MDS criteria for probable PD dementia). Conversion was defined as -1: conversion to a worse classification (ie, NC to MCI, NC to dementia or MCI to dementia), 0: no change, or 1: conversion to a better classification (ie, dementia to NC, MCI to NC, dementia to MCI).
Time Frame: One year after completion of the intervention (T3)
Population: Healthy control subjects did not undergo follow-up assessments. Number of participants analyzed differs from total population due to drop-out and missed assessment.
Measure: Number; unit: participants
Arm/Group | Online Cognitive Training 1 (N=68) | Online Cognitive Training 2 (N=68)
Number analyzed (Participants) | 56 | 53
participants
  -1: Conversion to worse classification | 12 | 11
  0: No change | 28 | 27
  1: Conversion to better classification | 16 | 15

10. Secondary Outcome: Performance on the Stroop Color-Word Test, Card I
Description: Processing speed change after eight weeks of cognitive training, measured with the Stroop Color Word Test (word-reading), where a higher time to completion indicates worse cognitive function.
Time Frame: Baseline (T0, "Pre-intervention") to eight weeks (T1, "Post-intervention")
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2 | Healthy Control Subjects
Number analyzed (Participants) | 67 | 66 | 29
time in seconds
  Baseline (T0) | 54.1 (10.7) | 56.3 (15.1) | 49.2 (9.4)
  Eight weeks (T1): number analyzed (Participants) | 67 | 66 | 0
  Eight weeks (T1) | 50.8 (9.1) | 54.3 (13.2) |

11. Secondary Outcome: Performance on the Stroop Color-Word Test, Card III
Description: Executive function CHANGE after eight weeks of cognitive training, measured with the Stroop Color Word Test (card III, color-word interference), where a higher time to completion indicates worse cognitive function.
Time Frame: Baseline (T0, "Pre-intervention") to eight weeks (T1, "Post-intervention")
Population: Three participants dropped out of the study and did not perform the T1 measurement and one participant did not undergo card III of the Stroop color word test at T1; these participants were subsequently removed from analyses. Healthy control subjects did not perform the second assessment.
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | Online Cognitive Training 1 | Online Cognitive Training 2 | Healthy Control Subjects
Number analyzed (Participants) | 67 | 65 | 29
time in seconds
  Baseline (T0) | 114.9 (49.3) | 106.9 (33.9) | 85.9 (19.0)
  Eight weeks (T1): number analyzed (Participants) | 67 | 65 | 0
  Eight weeks (T1) | 101.7 (28.6) | 103.4 (30.7) |

12. Secondary Outcome: Conversion of Cognitive Status at Two-year Follow-up
Description: Count of conversion of cognitive status at two-year follow-up with respect to the cognitive status at baseline (T0). Cognitive status is defined as cognitively normal (NC), mild cognitive impairment (MCI, according to cognitive aspects of level II MDS criteria), or dementia (according to cognitive aspects of MDS criteria for probable PD dementia). Conversion was defined as -1: conversion to a worse classification (ie, NC to MCI, NC to dementia or MCI to dementia), 0: no change, or 1: conversion to a better classification (ie, dementia to NC, MCI to NC, dementia to MCI).
Time Frame: Two year after completion of the intervention (T3)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Online Cognitive Training 1 (N=68) | Online Cognitive Training 2 (N=68)
Number analyzed (Participants) | 53 | 51
participants
  -1: Conversion to worse classification | 13 | 14
  0: No change | 25 | 27
  1: Conversion to better classification | 15 | 10

13. Other Pre Specified Outcome: Difference Between Parkinson's Disease Patients' Brain Network Topology With or Without Cognitive Impairment, and Healthy Control Subjects.
Description: Participants will be classified to cognitive impairment or no cognitive impairment, and their brain network topology will be compared with healthy subjects.
Time Frame: Pre-intervention (T0)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Online Cognitive Training Effect on Brain Network Topology Relative to Healthy Control Group
Description: The effect of online cognitive training on brain network topology using resting state fMRI compared with brain network topology of healthy subjects. Healthy subjects will undergo (functional) MRI scanning once.
Time Frame: Eight weeks (T1)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Online Cognitive Training Effect on Brain Activity Measured by Resting State fMRI
Description: The effect of online cognitive training on brain activity using resting state fMRI. Regional activity and functional connectivity changes will be assessed after eight weeks of training (T1).
Time Frame: Eight weeks (T1)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Online Cognitive Training Effect on Structural Brain Connectivity Measured by DTI
Description: The effect of online cognitive training on structural brain connectivity using DTI. Structural changes will be assessed after eight weeks of training (T1).
Time Frame: Eight weeks (T1)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Online Cognitive Training Effect on Brain Morphology Measured by MRI
Description: The effect of online cognitive training on brain morphology using MRI. Structural changes will be assessed after eight weeks of training (T1).
Time Frame: Eight weeks (T1)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Age
Description: Demographic characteristic: age at baseline.
Time Frame: Pre-intervention (T0)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Sex
Description: Demographic characteristic: sex.
Time Frame: Pre-intervention (T0)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Educational Level
Description: Demographic characteristic: educational level.
Time Frame: Pre-intervention (T0)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Disease Duration
Description: Disease characteristic: disease duration.
Time Frame: Pre-intervention (T0)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Disease Stage
Description: Disease characteristic: disease stage (Hoehn and Yahr stage).
Time Frame: Pre-intervention (T0), one year (T3), two years (T4)
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Medication Use
Description: Disease characteristic: medication use.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Motor Symptoms
Description: Motor symptoms assessed by the Unified Parkinson's Disease Rating Scale - III
Time Frame: Pre-intervention (T0), one year (T3), two years (T4)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Depressive Symptom Severity
Description: Psychiatric symptom severity, depression (Beck Depression Inventory).
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Anxiety Symptom Severity
Description: Psychiatric symptom severity, including anxiety (Parkinson Anxiety Scale).
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Impulse Control Disorder Symptom Severity
Description: Psychiatric symptom severity, including impulse control disorders (QUIP-RS).
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Psychotic Symptom Severity
Description: Psychiatric symptom severity, including psychotic symptoms (Questionnaire for psychotic events).
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Apathy Symptom Severity
Description: Psychiatric symptom severity, including apathy (Apathy Scale).
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Expectations of the Intervention
Description: Participants' expectation prior the intervention, measured by the credibility/expectancy questionnaire.
Time Frame: Pre-intervention (T0)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Global Cognitive Functioning (1)
Description: Global cognitive functioning assessed by the Montreal Cognitive Assessment (MoCA).
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Global Cognitive Functioning (2)
Description: Global cognitive functioning assessed by the Pentagon copy test, which is predictive of cognitive deterioration.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Specific Cognitive Functioning: Attention/Working Memory (1)
Description: Attention function, measured by the Stroop task part I: word naming.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Specific Cognitive Functioning: Attention/Working Memory (2)
Description: Working memory function, measured by the backwards digit span test of the Wechsler adult intelligence test (WAIS)-III.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Specific Cognitive Functioning: Episodic Memory (1)
Description: Episodic memory function, measured by the Dutch version of the Auditory verbal learning test (RAVLT).
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Specific Cognitive Functioning: Episodic Memory (2)
Description: Episodic memory function, measured by the Location learning task.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Specific Cognitive Functioning: Language (1)
Description: Language function, measured by the Boston naming task.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Specific Cognitive Functioning: Language (2)
Description: Language function, measured by the category fluency task.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Specific Cognitive Functioning: Visuospatial/Visuoconstructive Function (1)
Description: Visuospatial function, measured by the Benton visual form discrimination task.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Specific Cognitive Functioning: Visuospatial/Visuoconstructive Function (2)
Description: Visuospatial function, measured by the Rey complex figure task.
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Physical Activity
Description: Amount of estimated physical activity that a person performs, measured by the New Zealand Physical Activity Questionnaire
Time Frame: Pre-intervention (T0), eight weeks (T1), six months (T2), one year (T3), two years (T4)
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Cognitive Reserve
Description: Estimation of cognitive reserve measured with the Cognitive Reserve Index questionnaire
Time Frame: Two years (T4)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years (duration of study)
Description: No serious adverse events related to the intervention were expected due to the non-pharmacological nature of the intervention. We did collect information on the development of impulse control disorders to gain information about the risk of developing internet/gaming addiction as a result of cognitive training.
  Adverse events were logged.
Arm/Group | Online Cognitive Training 1 (N=68) | Online Cognitive Training 2 (N=68) | Healthy Control Subjects (N=31)
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/68 | 0/31
Other Adverse Events (participants affected / at risk) | 9/68 | 10/68 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Online Cognitive Training 1 (N=68) (N=68) | Online Cognitive Training 2 (N=68) (N=68) | Healthy Control Subjects (N=31) (N=31)
Impulse control disorder (Psychiatric disorders) | 0 | 1 (1) | 0 (0) — Development of punding during the study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Online Cognitive Training 1 (N=68) (N=68) | Online Cognitive Training 2 (N=68) (N=68) | Healthy Control Subjects (N=31) (N=31)
Medical issue related to PD (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) — Medical symptoms related to PD
Training-related adverse event (General disorders) | 3 (3) | 0 (0) | 0 (0) — Stress due to intervention
Medical issue not PD-related: COVID (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — COVID infection
Medical issue other than PD: Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Ear infection
Medical issue other than PD: injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) — Injury due to accident
Medical issue other than PD: meningioma (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) — Complications due to meningioma
Medical issue other than PD: cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) — Cerebral infarction
Medical issue other than PD: Restless legs and hyperventilation (General disorders) | 1 (1) | 0 (0) | 0 (0) — Restless legs and hyperventilation
Medical issue other than PD: dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0) — Dizziness

LIMITATIONS AND CAVEATS:
Sample size fell short of the intended statistical power: the initial sample size calculation was based on a within-between interaction of a repeated-measures ANOVA (corrected for pre-post assessment correlation r=.6) based on an effect size f=0.12 of CT on global cognitive function (Leung et al 2015). After trial completion we discovered this sample size is insufficient to detect the expected effect on global cognition due to obscurity in effect size parameter definition in G*Power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT02920632/Prot_SAP_000.pdf